CLINICAL TRIAL: NCT03541603
Title: A Double-Blind, Randomized, Placebo-Controlled Study of Levosimendan in Pulmonary Hypertension Patients With Heart Failure With Preserved Left Ventricular Ejection Fraction (PH-HFpEF)
Brief Title: Hemodynamic Evaluation of Levosimendan in Patients With PH-HFpEF
Acronym: HELP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tenax Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TNX-LVO-04
Record Dates: First submitted 2018-05-03; First posted 2018-05-30 (Actual); Results first posted 2024-05-14 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2020-04

CONDITIONS: Hypertension Pulmonary Secondary; Heart Failure, Right Sided; Heart Failure With Normal Ejection Fraction
Keywords: PH-HFpEF
MeSH Terms: conditions — Heart Failure | interventions — Simendan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Levosimendan 2.5mg/mL Injectable Solution (Experimental): 0.075 - 0.1µg/kg/min for 24 hrs (weekly)
  Interventions: Drug: Levosimendan
- Matching Placebo (Placebo Comparator): 0.075 - 0.1µg/kg/min for 24 hrs (weekly)
  Interventions: Drug: Matching Placebo

INTERVENTIONS:
Drug: Levosimendan — A sterile 2.5 mg/mL concentrate solution that is diluted in 5% Dextrose or 0.9 Normal Saline to achieve a 50 microgram/min solution for infusion
  Other Names: Levosimendan 2.5 mg/mL Injectable Solution
  Arms: Levosimendan 2.5mg/mL Injectable Solution
Drug: Matching Placebo — A sterile 2.5mg/mL concentrate solution that is diluted in 5% Dextrose or 0.9 Normal Saline to achieve a 50 microgram/min solution for infusion
  Other Names: Placebo
  Arms: Matching Placebo

SUMMARY:
Phase 2 study to evaluate the efficacy and safety of intermittent levosimendan compared with placebo in hemodynamic improvement with exercise in PH-HFpEF subjects

DETAILED DESCRIPTION:
Levosimendan and its prolonged active metabolite, OR-1896, have been shown to have favorable hemodynamic effects in subjects with pulmonary hypertension and right heart failure. Clinical studies that have been conducted in subjects with right heart failure and pulmonary hypertension suggest levosimendan may be an effective therapy in treatment of subjects with PH-HFpEF. This study will provide demonstration of levosimendan/OR-1896's effectiveness in critical measures of hemodynamic response in weekly administration of levosimendan and the concomitant response as measured by exercise capacity, subject quality of life, and changes in functional capacity. These data will support and guide the Phase 3 development of levosimendan in PH-HFpEF subjects.

ELIGIBILITY:
Inclusion Criteria:

Criteria to enter Open-label, Lead-in Dose Phase:

* Diagnosis of World Health Organization (WHO) Group 2 Pulmonary Hypertension (PH) with Heart Failure with Preserved Ejection Fraction (HFpEF) confirmed at the time of the diagnosis of pulmonary hypertension.
* Baseline Pulmonary Arterial Pressure (PAP) ≥35, Pulmonary Capillary Wedge Pressure (PCWP) ≥20, New York Heart Association (NYHA) Class IIb/III, Left Ventricular Ejection Fraction (LVEF) ≥40%
* Ability to walk at least 50 meters, but not more than 550 meters in a six-minute walk test.
* Stable oxygen treatment (if applicable), and medications for heart failure, hypertension, and respiratory condition

Criterion for Randomization to Double-blind Phase:

* Response to Open-label, Lead-in Levosimendan: Patients who demonstrate a ≥4mmHg reduction in PCWP from baseline measured at bicycle exercise (25 watts) with no more than a 10% decrease from baseline in cardiac index

Exclusion Criteria:

* Subject has a primary diagnosis of PH other than Group 2 PH-HFpEF
* Previous Percutaneous Coronary Intervention (PCI) or cardiac surgery (CABG), unless they have a negative stress test in the last 12 months)
* Congenital heart disease
* Clinically significant lung disease
* Planned heart or lung surgery
* Cardiac Index >4.0 L/min/m2
* Concomitant administration of pulmonary vasodilator therapy or taken within 14 days
* Dialysis or Glomerular Filtration Rate (GFR) <30 mL/min/1.73 m2
* Liver dysfunction with Child-Pugh Class B or C
* Evidence of systemic infection
* Weight > 150kg
* Symptomatic systolic blood pressure (SBP) cannot be managed to ensure SBP >100 mmHg
* Heart rate >= 100 bpm with the study drug, symptomatic and persistent for at least 10 minutes
* Hemoglobin < 80 g/L
* Serum potassium < 3.0 mmol/L or > 5.5 mmol/L at baseline
* Patients having severely compromised immune function
* Pregnant, suspected to be pregnant, or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2018-11-14 (Actual); Primary Completion 2020-04-07 (Actual); Study Completion 2020-04-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (16):
- United States (16):
  - Stanford Healthcare, Stanford, California
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Tufts Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - University of Minnesota Medical Center, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - University of Nebraska Medical Center, Omaha, Nebraska
  - North Shore University Hospital, Manhasset, New York
  - New York Presbyterian Hospital-Weill Cornell Medicine, New York, New York
  - Ichan School of Medicine at Mount Sinai, New York, New York
  - Christ Hospital, Cincinnati, Ohio
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh Presbyterian Hospital, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - UW Health University Hospital, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Burkhoff D, Rich S, Pollesello P, Papp Z. Levosimendan-induced venodilation is mediated by opening of potassium channels. ESC Heart Fail. 2021 Dec;8(6):4454-4464. doi: 10.1002/ehf2.13669. Epub 2021 Oct 30. PMID 34716759
- [Derived] Burkhoff D, Borlaug BA, Shah SJ, Zolty R, Tedford RJ, Thenappan T, Zamanian RT, Mazurek JA, Rich JD, Simon MA, Chung ES, Raza F, Majure DT, Lewis GD, Preston IR, Rich S. Levosimendan Improves Hemodynamics and Exercise Tolerance in PH-HFpEF: Results of the Randomized Placebo-Controlled HELP Trial. JACC Heart Fail. 2021 May;9(5):360-370. doi: 10.1016/j.jchf.2021.01.015. Epub 2021 Apr 7. PMID 33839076

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 44 patients satisfied entry criteria for enrollment and received lead-in open-label levosimendan.
  37 of the 44 enrolled patients achieved responder criteria following 24hr lead-in open label levosimendan infusion and were randomized to study
Period: Overall Study
Arm/Group | Levosimendan 2.5mg/mL Injectable Solution | Matching Placebo
Started | 18 | 19
Completed | 18 | 17
Not Completed | 0 | 2

BASELINE CHARACTERISTICS:
Population: One placebo patient failed to complete 6 weeks on study and was replaced as per protocol.
  One placebo patient was not able to return for Week 6 visit due to COVID-19 scheduling
Groups:
- Total: Total of all reporting groups
Arm/Group | Levosimendan 2.5mg/mL Injectable Solution | Matching Placebo | Total
Number analyzed (Participants) | 18 | 19 | 37
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.8 (7.5) | 67.4 (11.0) | 68.1 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 12 | 22
  Male | 8 | 7 | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 16 | 17 | 33
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 18 | 19 | 37

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline Pulmonary Capillary Wedge Pressure (PCWP) With Bicycle Exercise
Description: Change from baseline Pulmonary Capillary Wedge Pressure (PCWP) with bicycle exercise at Week 6
Time Frame: Baseline, Week 6
Population: patients completing Baseline and Week 6 visit with hemodynamic data
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Levosimendan 2.5mg/mL Injectable Solution | Matching Placebo
Number analyzed (Participants) | 18 | 17
mmHg | -1.9 (10.07) | -0.5 (7.87)

2. Secondary Outcome: Change in Cardiac Index (CI) at Rest and With Exercise.
Description: Change in Cardiac Index (CI) at rest and with exercise at Week 6 (CI determined by thermodilution) (CI is a hemodynamic parameter that relates the cardiac output (CO) from left ventricle in one minute to body surface area (BSA))
Time Frame: Baseline, Week 6
Population: patients completing Baseline and Week 6 visit with hemodynamic data
Measure: Mean (Standard Deviation); unit: L/min/m^2
Arm/Group | Levosimendan 2.5mg/mL Injectable Solution | Matching Placebo
Number analyzed (Participants) | 18 | 17
L/min/m^2
  rest | 0.05 (0.699) | -0.15 (0.262)
  exercise | 0.24 (1.106) | 0.04 (0.594)

3. Secondary Outcome: Change in Pulmonary Vascular Resistance (PVR) Effect at Rest and With Exercise
Description: Change in Pulmonary Vascular Resistance (PVR) effect at rest and with exercise at Week 6
Time Frame: Baseline, Week 6
Population: patients completing Baseline and Week 6 visit with hemodynamic data
Measure: Mean (Standard Deviation); unit: mmHg.min/L
Arm/Group | Levosimendan 2.5mg/mL Injectable Solution | Matching Placebo
Number analyzed (Participants) | 18 | 17
mmHg.min/L
  rest | -0.09 (1.050) | 0.15 (2.238)
  exercise | -0.44 (1.539) | -0.16 (1.81)

4. Secondary Outcome: Change in PCWP When Supine and Legs Elevated
Description: Change in Pulmonary Capillary Wedge Pressure, Baseline to Week 6
Time Frame: Baseline, Week 6
Population: patients completing Baseline and Week 6 visit with hemodynamic data
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Levosimendan 2.5mg/mL Injectable Solution | Matching Placebo
Number analyzed (Participants) | 18 | 17
mmHg
  rest | -5.1 (5.26) | -1.7 (6.14)
  legs elevated | -6.0 (7.75) | -0.3 (5.45)

5. Secondary Outcome: Patient Global Assessment
Description: Patient assessment of well-being based on 6 questions assessed on a 5-point Likert Scale ( 1 =worst, 5= best) (minimum total score 5pts, maximum total score 25 pts) (no comparison to baseline as no instrument used at baseline)
Time Frame: Baseline, Week 6
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Levosimendan 2.5mg/mL Injectable Solution | Matching Placebo
Number analyzed (Participants) | 18 | 17
units on a scale | 3 [3 to 4] | 3 [3 to 4]

6. Secondary Outcome: Exercise Duration Via 6 Minute Walk Test
Description: Change in 6-minute walk test at Week 6 vs baseline
Time Frame: Baseline, Week 6
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Levosimendan 2.5mg/mL Injectable Solution | Matching Placebo
Number analyzed (Participants) | 18 | 17
meters | 16.6 (40.03) | -12.8 (35.08)

7. Secondary Outcome: Physician's Assessment of Functional Class
Description: Physician's Assessment of New York Heart Association (NYHA) Classification (one of four categories based on how much the patient is limited during physical activity. (Class I, no limitation of physical activity to Class IV, marked limitation of physical activity).
Time Frame: Baseline, Week 6
Measure: Count of Participants; unit: Participants
Arm/Group | Levosimendan 2.5mg/mL Injectable Solution | Matching Placebo
Number analyzed (Participants) | 18 | 17
Participants
  Baseline: Class I | 0 | 0
  Baseline: Class II | 2 | 3
  Baseline: Class III | 16 | 14
  Baseline: Class IV | 0 | 0
  Week 6: Class I | 0 | 0
  Week 6: Class II | 8 | 5
  Week 6: Class III | 10 | 12
  Week 6: Class IV | 0 | 0

8. Secondary Outcome: Number of Participants With Composite Events of Death or Hospitalization
Description: Number of Participants with Composite Events of death or hospitalization through Week 6
Time Frame: Baseline, Week 6
Measure: Count of Participants; unit: Participants
Arm/Group | Levosimendan 2.5mg/mL Injectable Solution | Matching Placebo
Number analyzed (Participants) | 18 | 17
Participants | 3 | 1

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | Levosimendan 2.5mg/mL Injectable Solution | Matching Placebo
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/19
Serious Adverse Events (participants affected / at risk) | 3/18 | 1/19
Other Adverse Events (participants affected / at risk) | 13/18 | 8/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Levosimendan 2.5mg/mL Injectable Solution (N=18) | Matching Placebo (N=19)
Device related infection (Infections and infestations) | 1 (1) | 0 (0) — PICC LINE INFECTION WITH DUE TO Serious Adverse Event (SAE) associated with Peripherally Inserted Central Venous Catheter (PICC) HOSPITALIZATION
Bacteremia (Infections and infestations) | 1 (1) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 2 (2) | 0 (0)
Cardiogenic Shock (Cardiac disorders) | 0 (0) | 1 (1)
Right ventricular failure (Cardiac disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Levosimendan 2.5mg/mL Injectable Solution (N=18) | Matching Placebo (N=19)
Fatigue (General disorders) | 1 (1) | 2 (2)
Chills (General disorders) | 1 (1) | 1 (1)
Infusion site hemorrhage (General disorders) | 1 (1) | 1 (1)
Infusion site erythema (General disorders) | 1 (1) | 0 (0)
Edema (General disorders) | 1 (1) | 0 (0)
Peripheral swelling (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 2 (2) | 1 (1)
Cardiogenic shock (Cardiac disorders) | 0 (0) | 1 (1)
Extrasystoles (Cardiac disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Right ventricular failure (Cardiac disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 1 (1)
Atypical pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Bacteremia (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis viral (Infections and infestations) | 0 (0) | 1 (1)
Device-related infection (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Tooth abscess (Infections and infestations) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 3 (3) | 1 (1)
Balance disorder (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness postural (Nervous system disorders) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Vascular access site pain (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Accidental overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Underdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Heart rate increased (Investigations) | 2 (2) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0)
Body temperature increased (Investigations) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Device infusion issue (Product Issues) | 1 (1) | 1 (1)
Device dislocation (Product Issues) | 1 (1) | 0 (0)
Device occlusion (Product Issues) | 0 (0) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Lactic acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin necrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Peripheral artery stenosis (Vascular disorders) | 0 (0) | 1 (1)
Thrombophlebitis (Vascular disorders) | 1 (1) | 0 (0)
Venous thrombosis limb (Vascular disorders) | 1 (1) | 0 (0)
Vison blurred (Eye disorders) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Hemodynamic effects at Wk6 were measured ~1 week after final levosimendan infusion. Thus, hemodynamic effects at 6 weeks represent effects at trough levels; greater effects might have been observed with earlier assessment.

No previous study evaluated chronic levosimendan in PH-HFpEF. Chose a low dose out of an abundance of caution. It remains possible that higher doses may be more effective in selected patients.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-05-15): https://cdn.clinicaltrials.gov/large-docs/03/NCT03541603/Prot_000.pdf
  • Statistical Analysis Plan (2019-05-18): https://cdn.clinicaltrials.gov/large-docs/03/NCT03541603/SAP_001.pdf